CLINICAL TRIAL: NCT03285516
Title: Improving Access to Evidence Based Care Among Rural Veterans Using a Transdiagnostic Treatment Approach
Brief Title: Safety Aid Reduction Treatment for Rural Veterans
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Collaborators: South Central Mental Illness Research Education and Clinical Center (Unknown)
Responsible Party: Principal Investigator, C Laurel Franklin, PhD, Clinical Psychologist, Southeast Louisiana Veterans Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 351
Record Dates: First submitted 2017-07-12; First posted 2017-09-18 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Emotional Disorder
Keywords: transdiagnostic treatment; emotional disorders; veterans; rural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- START (Experimental): The Safety Aid Reduction Treatment (START) protocol will consist of eight group sessions, delivered once weekly, lasting approximately one hour in duration. START will be delivered in-person by the PI and group co-leader.
  Interventions: Behavioral: Safety Aid Reduction Treatment

INTERVENTIONS:
Behavioral: Safety Aid Reduction Treatment — START includes many of the key elements found in empirically supported treatments for emotional disorders including a) psychoeducation regarding the nature of distress and b) exposure to internal sensations and external situations that are connected to one's distress response via identification and reduction in safety aids. Safety aids discussed in the current protocol include cognitive avoidance, situational avoidance, checking behaviors, reassurance seeking, avoidance of bodily sensations, companions, and use of alcohol and other substances.

SUMMARY:
The primary aim of the current proposal is to test the acceptability and feasibility of a group-based transdiagnostic treatment, termed Safety Aid Reduction Treatment (START), delivered to rural Veterans. The anticipated results of the proposed study include: 1) START will be both acceptable and feasible to Veterans and mental health care providers, alike and 2) START will lead to meaningful reductions in symptoms of anxiety and depression.

DETAILED DESCRIPTION:
This is an intervention pilot project examining the acceptability, feasibility, and utility of a group-based transdiagnostic treatment delivered to rural Veterans. Approximately 5.2 million Veterans reside in rural communities across the United States, making it difficult for them to access quality medical and mental health (MH) care. The Department of Veterans Affairs (VA) established Community Based Outpatient Clinics (CBOCs) to improve access to healthcare for rural Veterans; however, these clinics often lack MH specialists including psychiatrists and psychologists, limiting the breadth of specialty services available. As such, MH care is often delivered by primary care providers or MH clinicians who (a) lack familiarity with evidence-based interventions and (b) lack the time needed to implement such intensive therapies. Group-based cognitive behavioral protocols that target a number of different diagnoses are likely to be more attractive in these settings and therefore more readily disseminated. Such protocols, often referred to as transdiagnostic treatments, are based on the theory that emotional disorders share common features and therefore respond to common therapeutic procedures. One such treatment, termed Safety Aid Reduction Treatment (START), has received increasing empirical support. This group-based transdiagnostic treatment is designed to address cognitive and behavioral strategies, otherwise known as safety aids, that are common across a number of psychiatric conditions (e.g., anxiety disorders, trauma- and stressor-related disorders, obsessive-compulsive and related disorders, and depressive disorders) and used to reduce anxiety. START has been found to effectively reduce psychopathology in community-based clinical samples and more recently among Veterans at the Southeast Louisiana Veterans Health Care System (SLVHCS). However, the utility of this treatment has yet to be examined in rural settings. Thus, the primary aim of the current proposal is to test the acceptability and feasibility of a group-based transdiagnostic treatment, termed START, delivered to rural Veterans at CBOCs. Because this is a pilot project, we will not emphasize symptom reduction, as we will likely be underpowered to detect treatment effects. Nevertheless, a secondary aim of the project is to examine the utility of START by gathering data on symptom change, which will be used as pilot data for a subsequent grant proposal. For this pilot project, Veterans (N = 24) will be recruited from two of the five Southeast Louisiana Veterans Health Care System (SLVHCS) CBOCs. The anticipated results of the proposed study include: 1) START will be both acceptable and feasible to Veterans and mental health care providers, alike and 2) START will lead to meaningful reductions in symptoms of anxiety and depression. Findings from the current study will help to advance our understanding of the amelioration of anxiety and depressive disorders among Veterans.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Veterans must be diagnosed with an emotional disorder (e.g., anxiety disorder, obsessive-compulsive and related disorder, trauma-and stressor-related disorder, depressive disorder).
* And be primarily served at a CBOC location.

Exclusion Criteria:

* < 18 years of age
* Currently dependent upon substances and in need of detoxification
* Evidence of active psychosis
* Acutely suicidal or homicidal
* Uncontrolled bipolar disorder (e.g., not stable on medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
START Qualitative Treatment Questionnaire | 8 weeks
  The START Qualitative Treatment Questionnaire is a brief, structured short-answer qualitative questionnaire that was developed by the research team to assess Veterans experience with the START protocol.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) | Baseline and 8 weeks and 12 weeks
  The OASIS is a brief 5-item self-report questionnaire that can be used to assess anxiety severity and impairment across a number of anxiety diagnoses. Participants will be asked to respond to items regarding their experience with anxiety and fear over the past week using a zero (No anxiety) to four (Constant anxiety) Likert-type scale. Items are summed to create a total score with higher scores indicating greater anxiety severity.
Overall Depression Severity and Impairment Scale (ODSIS) | Baseline and 8 weeks and 12 weeks
  The ODSIS is a brief 5-item self-report questionnaire that can be used to assess depression severity and impairment across heterogeneous mood disorders. Participants will be asked to respond to items regarding their experience with depression over the past week using a zero (No depression) to four (Constant depression) Likert-type scale. Items are summed to create a total score with higher scores indicating greater depression severity.
Safety Behavior Assessment Form (SBAF) | Baseline and 8 weeks and 12 weeks
  The SBAF is a 41-item self-report questionnaire designed to assess safety behavior usage. Participants will be asked to read a list of behaviors that people sometimes use to make themselves feel more comfortable and pick the response that most accurately describes how often they engage in that behavior using a zero (Never) to three (Always) Likert-type scale. Items are summed to create a total score with higher scores indicating greater safety aid usage.
Work and Social Adjustment Scale (WSAS) | Baseline and 8 weeks and 12 weeks
  The WSAS is a 5-item descriptive measure of subjective interference of psychiatric symptoms in various life domains (i.e., work, home, leisure, and family). Participants will be asked to read a list of problems and determine how much the problem impairs their ability to carry out the activity using a zero (Not at all) to eight (Very severely) Likert-type scale. Items are summed to create a total score with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M. Raines, Ph.D., Principal Investigator — Southeast Louisiana Veterans Health Care System
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Data sets underlying this project will not be shared outside the VA, except as required under the Freedom of Information Act (FOIA), for a number of reasons. First, data will be used by the research team to answer additional research questions. Further, veterans may be hesitant to participate in research in which the data will be shared outside the VA and this may act as a barrier to participation and/or benefit from treatment.

REFERENCES:
- [Background] Veterans Health Administration Office of Rural Health. ORH Fact Sheet. 2014; Available from: http://www.ruralhealth.va.gov.
- [Background] Allen, L.B., R.K. McHugh, and D.H. Barlow, Emotional disorders: A unified protocol. 2008.
- [Background] Schmidt NB, Buckner JD, Pusser A, Woolaway-Bickel K, Preston JL, Norr A. Randomized controlled trial of false safety behavior elimination therapy: a unified cognitive behavioral treatment for anxiety psychopathology. Behav Ther. 2012 Sep;43(3):518-32. doi: 10.1016/j.beth.2012.02.004. Epub 2012 Mar 9. PMID 22697441
- [Background] Riccardi CJ, Korte KJ, Schmidt NB. False Safety Behavior Elimination Therapy: A randomized study of a brief individual transdiagnostic treatment for anxiety disorders. J Anxiety Disord. 2017 Mar;46:35-45. doi: 10.1016/j.janxdis.2016.06.003. Epub 2016 Jun 18. PMID 27397584